CLINICAL TRIAL: NCT05924308
Title: Acupuncture Therapy for Post-stroke Mild Cognitive Impairment: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YD202219
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2022-09

CONDITIONS: Post-stroke Mild Cognitive Impairment
Keywords: Acupuncture therapy
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator)
  Interventions: Other: sham acupuncture
- treatment group (Experimental)
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — every time 30 min, 1 times a day, five times a week, 4 weeks for 1 course of treatment, treatment 3 period of treatment.
  Arms: treatment group
Other: sham acupuncture — Electroacupuncture was connected to the fixed place of Sishencong on the left and right sides of Baihui and Shenting, and the electroacupuncture instrument was returned to zero. Pull out the needle when informed patient for cotton on the above points, to make patients feel the needle was pulled out. The same treatment time of 30 min, 1 times a day, five times a week, 4 weeks for 1 course of treatment, treatment 3 period of treatment.
  Arms: control group

SUMMARY:
1. On the basis of previous studies, standardized randomized controlled clinical trials were conducted to observe the efficacy and safety of acupuncture in the treatment of mild cognitive impairment after stroke using the international rating scale, and the clinical experience was transformed into evidence.
2. According to the clinical outcomes reported by patients, the differences between Chinese and western scales in evaluating mild cognitive impairment after stroke were compared. On the basis of "disease differentiation, syndrome differentiation and meridian differentiation", the syndrome differentiation and treatment system of mild cognitive impairment after stroke was preliminarily constructed, and the TCM syndrome prediction model was improved.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria: ① Stroke diagnostic criteria: according to the diagnostic criteria of cerebral infarction and cerebral hemorrhage in the "Chinese Guidelines for the Prevention and Treatment of Stroke (2021 edition)" issued by the National Health Commission, the diagnosis was confirmed by head CT or MRI examination. ② Mild cognitive impairment diagnostic criteria: according to the 2018 Chinese Guidelines for the Diagnosis and Treatment of Dementia and cognitive Impairment (5) : Diagnosis and treatment of mild cognitive Impairment. ③ TCM diagnostic criteria: according to the "TCM Diagnostic Efficacy Criteria" issued by the State Administration of Traditional Chinese Medicine in 2012, the patients were diagnosed as dementia.
2. 40 years old ≤ age ≤75 years old, regardless of gender;
3. cognitive impairment occurred after stroke without other causes;
4. cognitive impairment within 6 months after stroke;
5. stable condition, clear consciousness, MoCA score < 26 points;
6. those who were willing to participate in the study and signed the "informed consent".

Exclusion Criteria:

* Brain CT or MRI showed other lesions unrelated to stroke, or severe brain atrophy or leukoaraiosis; (2) serious complications (myocardial infarction, heart failure, malignant tumor, severe infection, mental illness, severe depression, epilepsy, etc.);

  * with obvious hearing impairment, visual impairment, aphasia and other inability to cooperate in the physical evaluation; (4) pregnant or intended to pregnant women, lactating women; ⑤ intolerance to acupuncture; ⑥ bleeding tendency and poor coagulation function.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
MMSE | week (0,4,8,12,20)
  Mini-mental State Examination scale

SECONDARY OUTCOMES:
MoCA | week (0,4,8,12,20)
  Montreal Cognitive Assessment
MBI | week (0,4,8,12,20)
  Modified Barthel Index
SSTCM | week (0,4,8,12,20)
SS-QOL | week (0,4,8,12,20)

CONTACTS AND LOCATIONS:
Locations (1):
- Longhua Hospital, Shanghai university of TCM, Shanghai, Shanghai Municipality, China